CLINICAL TRIAL: NCT00661141
Title: A Phase IIa, Prospective, Randomized, Blinded, Intra-Subject Controlled, Single Dose, Dose Escalation Study of Antizol® for Mitigation of Acetaldehyde Related Toxicity in Human Subjects With Symptoms of Inborn Altered Ethanol Metabolism With Concomitant Ethanol Exposure
Brief Title: Phase IIa Study of Fomepizole for Acetaldehyde Toxicity After Ethanol Exposure in Subjects With Altered Ethanol Metabolism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BP1-01-01
Record Dates: First submitted 2008-04-16; First posted 2008-04-18 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Aldehyde Dehydrogenase-2 (ALDH2) Deficiency
Keywords: acetaldehyde; ethanol; ALDH2
MeSH Terms: interventions — Fomepizole; 4-methylpiperazine-2,6-dione; Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1: Antizol 1.0 mg/kg (Experimental): Participants receive alternating study treatment (oral fomepizole 1.0 mg/kg or placebo) on 2 sequential days (Study Day 1 and Study Day 2), administered 30 minutes prior to ethanol or 30 minutes after ethanol.
  Interventions: Drug: Antizol; Drug: Placebo; Other: Ethanol
- Cohort 2: Antizol 3.0 mg/kg (Experimental): Participants receive alternating study treatment (oral fomepizole 3.0 mg/kg or placebo) on 2 sequential days (Study Day 1 and Study Day 2), administered 30 minutes prior to ethanol or 30 minutes after ethanol.
  Interventions: Drug: Antizol; Drug: Placebo; Other: Ethanol
- Cohort 3: Antizol 5.0 mg/kg (Experimental): Participants receive alternating study treatment (oral fomepizole 5.0 mg/kg or placebo) on 2 sequential days (Study Day 1 and Study Day 2), administered 30 minutes prior to ethanol.
  Interventions: Drug: Antizol; Drug: Placebo; Other: Ethanol
- Cohort 4: Antizol 1.0 mg/kg (Experimental): Participants receive alternating study treatment (oral fomepizole 7.0 mg/kg or placebo) on 2 sequential days (Study Day 1 and Study Day 2), administered 30 minutes prior to ethanol.
  Interventions: Drug: Antizol; Drug: Placebo; Other: Ethanol

INTERVENTIONS:
Drug: Antizol
  Other Names: fomepizole; 4-methylpyrazole; 4-MP
Drug: Placebo
Other: Ethanol — oral dose of ethanol (0.5 g/kg)

SUMMARY:
This trial will evaluate if fomepizole (4-methylpyrazole) can treat symptoms associated with alcohol intolerance due to aldehyde dehydrogenase 2 (ALDH2) deficiency, an inherited metabolic disorder. These symptoms include flushing, nausea, headache, shortness of breath and dizziness, resulting from exposure to acetaldehyde, the primary metabolite of ethanol. Long-term, serious health risks have been associated with repeated exposure to acetaldehyde, a carcinogen, among ALDH2-deficient individuals.

DETAILED DESCRIPTION:
Approximately 32 subjects will be enrolled in ascending dosing cohorts of 8 subjects each. Each subject will receive an oral dose of study drug (fomepizole or placebo) with concomitant ethanol with group assignment in a randomized 1:1:1:1 ratio (2 subjects each group) on Study Day 1. Each subject is their own intra-subject control with the alternative study drug (fomepizole or placebo) administered on the next day (Study Day 2). Four subjects in each cohort will receive study drug (fomepizole or placebo) administered 30 minutes prior to ethanol, 4 with study drug (fomepizole or placebo) administered 30 minutes after ethanol. The study will assess safety and tolerability of fomepizole and the PK/PD of 4-MP, ethanol and acetaldehyde in the subject population.

Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age 21 to 50 years
* Subject of Japanese descent
* History of flushing, with or without palpitations, or nausea (Alcohol Sensitivity Screening Test ≥ 3.1) following occasional or inadvertent ethanol consumption either currently or in the past
* Subjects must be healthy volunteers with no other clinically relevant abnormalities as determined by medical history, blood chemistry, complete blood count (CBC), urinalysis,and 12-lead electrocardiogram (ECG)
* Positive skin ethanol patch test (100 μL of 70% ethanol on a lint pad applied to skin for 7 minutes results in an area of erythema)
* For Cohort 4, enrolled subjects were either homozygous or heterozygous for the ALDH2*2 genotype as assessed by genotyping at Screening

Exclusion Criteria:

* Vaccination within 2 weeks of Day 1
* Current respiratory disease or a past history of chronic respiratory disease, or current smoker within last six months
* Any one of the following Screening ECG findings:

  * QTc (Bazett) interval duration greater than 450 msec (male) or 470 msec (female), or
  * QRS interval greater than 120 msec, or
  * PR interval greater than 220 msec
* History or evidence of drug or alcohol abuse or regular consumption of more than 8 units of alcohol daily (1 unit = 300 mL beer, 1 glass wine, 1 measure spirit) or those who may have difficulty abstaining from non study alcohol during the 36 hours prior to dose administration and until completion of blood sampling on Day 7
* Subjects who have donated blood totalling more than 550 mL within the 3 months prior to Day 1
* Use of any prescription medication other than oral contraceptives during the 14 days prior to Day 1, unless approved by both the Principal Investigator (PI) and the Sponsor
* Inability to abstain from smoking any tobacco product from within prior to 2 hours of blood sampling to after 2 hours of blood sampling during the study period.
* Use of any over-the-counter product, herbal product, diet aid, hormone supplement, etc., within 14 days prior to Day 1 unless approved by both the PI and the Sponsor
* Chronic use of pain medications
* Administration of an investigational agent within the last 30 days (or within a period of less than 5 times the agent's half-life, whichever is longer) prior to Day 1
* Major surgery within 60 days prior to Day 1, or any planned surgery or medical procedure during the study period (through Day 7)
* Positive alcohol breath-test or Positive drug screen (e.g., opiates, barbiturates, cannabinoids, benzodiazepines, cocaine, amphetamines) during screening or at Day 0 Check-In
* Known hypersensitivity reaction to Antizol® or other pyrazoles, tomato juice
* Abnormal laboratory results, including:

  * WBC ≤3.5 × 109/L or neutrophil count ≤2.0 × 10^9/L
  * Hemoglobin <12.0 or >16.0 gm/dL
  * Creatinine ≥2 mg/dL
  * Total bilirubin ≥2 mg/dL
  * Alanine aminotransferase and/or aspartate aminotransferase ≥2 times the upper limit of normal
  * PaO2 ≤95% on room air by pulse oximetry
  * Urine dipstick positive for protein, blood, ketones, glucose or leukocyte esterase
* Any other clinically significant abnormal result for hematology, clinical chemistry, or urinalysis at screening or check-In
* Positive serum pregnancy test for females of childbearing potential
* Subject and/or partner unable or unwilling to use an effective form of barrier contraceptives during the course of the study and for 7 days after study drug administration.
* Cancer (excluding adequately treated basal cell carcinoma) within the last 5 years
* Significant past medical history of hepatic, renal, cardiovascular (including family history of prolonged QT syndrome), pulmonary, gastrointestinal, hematological, locomotor, immunologic, ophthalmologic, metabolic endocrine or other diseases; or any condition that in the opinion of the Investigator would complicate or compromise the study, or the well-being of the subject
* Any other reason, which in the opinion of the Principal Investigator, would prevent the subject from completing or following the study schedule

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Covance Honolulu CRU, Honolulu, Hawaii, United States

REFERENCES:
- [Background] Inoue K, Fukunaga M, Kiriyama T, Komura S. Accumulation of acetaldehyde in alcohol-sensitive Japanese: relation to ethanol and acetaldehyde oxidizing capacity. Alcohol Clin Exp Res. 1984 May-Jun;8(3):319-22. doi: 10.1111/j.1530-0277.1984.tb05519.x. PMID 6377951
- [Background] Inoue K, Kera Y, Kiriyama T, Komura S. Suppression of acetaldehyde accumulation by 4-methylpyrazole in alcohol-hypersensitive Japanese. Jpn J Pharmacol. 1985 May;38(1):43-8. doi: 10.1254/jjp.38.43. PMID 4021229
- [Background] Tardif R, Liu L, Raizenne M. Exhaled ethanol and acetaldehyde in human subjects exposed to low levels of ethanol. Inhal Toxicol. 2004 Apr;16(4):203-7. doi: 10.1080/08958370490277272. PMID 15204767
- [Background] Yokoyama T, Yokoyama A, Kato H, Tsujinaka T, Muto M, Omori T, Haneda T, Kumagai Y, Igaki H, Yokoyama M, Watanabe H, Yoshimizu H. Alcohol flushing, alcohol and aldehyde dehydrogenase genotypes, and risk for esophageal squamous cell carcinoma in Japanese men. Cancer Epidemiol Biomarkers Prev. 2003 Nov;12(11 Pt 1):1227-33. PMID 14652286

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although originally planned to receive Antizol 7.0 mg/kg, participants in Cohort 4 were dosed with study drug (Antizol or placebo) at 1.0 mg/kg,the same level dosed for the Cohort 1 participants. As a result, Cohorts 1 and 4 were combined together in the data summary and statistical analyses.
Groups:
- Antizol 1.0 mg/kg, Then Placebo: Participants received Antizol 1.0 mg/kg then placebo treatment on 2 sequential days (Study Day 1 and Study Day 2), administered 30 minutes prior to ethanol or 30 minutes after ethanol.
- Placebo, Then Antizol 1.0 mg/kg: Participants received placebo treatment then Antizol 1.0 mg/kg on 2 sequential days (Study Day 1 and Study Day 2), administered 30 minutes prior to ethanol or 30 minutes after ethanol.
- Antizol 3.0 mg/kg, Then Placebo: Participants received Antizol 3.0 mg/kg then placebo treatment on 2 sequential days (Study Day 1 and Study Day 2), administered 30 minutes prior to ethanol or 30 minutes after ethanol.
- Placebo, Then Antizol 3.0 mg/kg: Participants received placebo treatment then Antizol 3.0 mg/kg on 2 sequential days (Study Day 1 and Study Day 2), administered 30 minutes prior to ethanol or 30 minutes after ethanol.
- Antizol 5.0 mg/kg, Then Placebo: Participants received Antizol 5.0 mg/kg then placebo treatment on 2 sequential days (Study Day 1 and Study Day 2), administered 30 minutes prior to ethanol.
- Placebo, Then Antizol 5.0 mg/kg: Participants received placebo treatment then Antizol 5.0 mg/kg on 2 sequential days (Study Day 1 and Study Day 2), administered 30 minutes prior to ethanol.
Period: Overall Study
Arm/Group | Antizol 1.0 mg/kg, Then Placebo | Placebo, Then Antizol 1.0 mg/kg | Antizol 3.0 mg/kg, Then Placebo | Placebo, Then Antizol 3.0 mg/kg | Antizol 5.0 mg/kg, Then Placebo | Placebo, Then Antizol 5.0 mg/kg
Started | 8 | 8 | 4 | 4 | 4 | 4
Administered 30 Minutes Prior to Ethanol | 6 | 6 | 2 | 2 | 4 | 4
Administered 30 Minutes After Ethanol | 2 | 2 | 2 | 2 | 0 | 0
Completed | 8 | 8 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Antizol 1.0 mg/kg and Placebo: Participants received alternating study treatment (oral Antizol 1.0 mg/kg or placebo) on 2 sequential days (Study Day 1 and Study Day 2), administered 30 minutes prior to ethanol or 30 minutes after ethanol.
- Antizol 3.0 mg/kg and Placebo: Participants receive alternating study treatment (oral Antizol 3.0 mg/kg or placebo) on 2 sequential days (Study Day 1 and Study Day 2), administered 30 minutes prior to ethanol or 30 minutes after ethanol.
- Antizol 5.0 mg/kg and Placebo: Participants receive alternating study treatment (oral Antizol 5.0 mg/kg or placebo) on 2 sequential days (Study Day 1 and Study Day 2), administered 30 minutes prior to ethanol or 30 minutes after ethanol.
- Total: Total of all reporting groups
Arm/Group | Antizol 1.0 mg/kg and Placebo | Antizol 3.0 mg/kg and Placebo | Antizol 5.0 mg/kg and Placebo | Total
Number analyzed (Participants) | 16 | 8 | 8 | 32
Age, Continuous [Mean (Full Range); unit: years] | 38 [28 to 50] | 29 [22 to 44] | 34 [23 to 43] | 34 [22 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 5 | 14
  Male | 10 | 5 | 3 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic/Latino | 16 | 8 | 8 | 32
  Asian | 16 | 8 | 8 | 32
  Japanese Ancestry | 16 | 8 | 8 | 32
  Born in Japan | 10 | 7 | 8 | 25
  Not Born in Japan | 6 | 1 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs, and AEs Leading to Study Discontinuation
Description: AEs were collected to evaluate the safety and tolerability of oral Antizol with concomitant ethanol administration in particitpants with symptoms of acetaldehyde toxicity associated with altered ethanol metabolism. AE: any untoward medical event that occurs following the first administration of study medication until the study participant's last study visit, whether or not the event is considered drug related. SAE: an event that meets any of the following criteria: results in death; is life threatening; requires inpatient hospitalization or prolongation of an existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect in the offspring of an exposed subject; is medically significant or an important medical event as assessed by investigator or sponsor; is, in the opinion of the investigator, an important medical event.
Time Frame: Study Day 0 through Study Visit Day 7
Measure: Count of Participants; unit: Participants
Groups:
- Antizol 1.0 mg/kg: Participants received alternating study treatment (oral Antizol 1.0 mg/kg or placebo) on 2 sequential days (Study Day 1 and Study Day 2), administered 30 minutes prior to ethanol or 30 minutes after ethanol.
- Antizol 3.0 mg/kg: Participants received alternating study treatment (oral Antizol 3.0 mg/kg or placebo) on 2 sequential days (Study Day 1 and Study Day 2), administered 30 minutes prior to ethanol or 30 minutes after ethanol.
- Antizol 5.0 mg/kg: Participants received alternating study treatment (oral Antizol 5.0 mg/kg or placebo) on 2 sequential days (Study Day 1 and Study Day 2), administered 30 minutes prior to ethanol.
- Pooled Placebo: Participants received placebo on either Study Day 1 or Study Day 2, administered 30 minutes prior to, or after, ethanol.
- Overall: Participants received alternating study treatment (oral Antizol 1.0, 3.0, or 5.0 mg/kg or placebo) on 2 sequential days (Study Day 1 and Study Day 2), administered 30 minutes prior to ethanol.
Arm/Group | Antizol 1.0 mg/kg | Antizol 3.0 mg/kg | Antizol 5.0 mg/kg | Pooled Placebo | Overall
Number analyzed (Participants) | 16 | 8 | 8 | 32 | 32
Participants
  Any AE | 13 | 6 | 8 | 21 | 28
  Mild AE | 13 | 6 | 8 | 19 | 28
  Moderate AE | 2 | 0 | 0 | 5 | 7
  Severe AE | 0 | 0 | 0 | 0 | 0
  Life-Threatening/Disabling AE | 0 | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0 | 0
  Possibly or Probably Related AE | 13 | 6 | 5 | 18 | 27
  AE Leading to Study Discontinuation | 0 | 0 | 0 | 0 | 0
  Serious AE | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK) of 4-MP: Maximum Plasma Concentration (Cmax)
Time Frame: Days 1 and 2: prior to administration of 1st treatment (ethanol or study drug); 10, 20, and 30 min prior to administration of second treatment (study drug or ethanol); 40, 50, 60 min and 2, 3, 4, 5, 6, and 8 hr post administration of 1st treatment
Population: Modified Intent-to-Treat: participants who received any study medication or procedure and who received study assessments through Study Day 2.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 1.0 mg/kg Antizol Followed by Ethanol: 1.0 mg/kg Antizol followed by ethanol 30 minutes later
- Ethanol Followed by 1.0 mg/kg Antizol: Ethanol followed by 1.0 mg/kg Antizol 30 minutes later
- 3.0 mg/kg Antizol Followed by Ethanol: 3.0 mg/kg Antizol followed by ethanol 30 minutes later
- Ethanol Followed by 3.0 mg/kg Antizol: Ethanol followed by 3.0 mg/kg Antizol 30 minutes later
- 5.0 mg/kg Antizol Followed by Ethanol: 5.0 mg/kg Antizol followed by ethanol 30 minutes later
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 8
ng/mL | 2386 (625) | 1358 (359) | 5605 (1183) | 4680 (645) | 8623 (2674)

3. Secondary Outcome: PK of 4-MP: Dose-Normalized (DN) Cmax
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: (ng/mL)/mg
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 8
(ng/mL)/mg | 38.3 (15.9) | 18.9 (4.65) | 27.6 (3.05) | 28.0 (4.26) | 30.2 (11.0)
Statistical Analysis 1: Comparison: 1.0 mg/kg Antizol Followed by Ethanol vs Ethanol Followed by 1.0 mg/kg Antizol vs 3.0 mg/kg Antizol Followed by Ethanol vs Ethanol Followed by 3.0 mg/kg Antizol vs 5.0 mg/kg Antizol Followed by Ethanol; 1.0 mg/kg Cohort, 3.0 mg/kg cohort, 5.0 mg/kg cohort; Test type: Superiority; p = 0.8727, ANOVA — Overall p-value testing cohort difference from ANOVA

4. Secondary Outcome: PK of 4-MP: Time to Cmax (Tmax)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 8
hours | 1.00 [0.333 to 4.00] | 2.50 [1.53 to 4.43] | 0.667 [0.333 to 1.00] | 1.48 [0.500 to 2.50] | 1.00 [0.333 to 3.00]

5. Secondary Outcome: PK of 4-MP: Area Under the Plasma Concentration-Time Curve (AUC), Calculated to the Last Measured Concentration (AUC[0-t])
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 8
ng*hr/mL | 13804 (4492) | 7409 (1437) | 44942 (17784) | 34310 (14431) | 109298 (30635)

6. Secondary Outcome: PK of 4-MP: DN AUC(0-t)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: (ng*hr/mL)/mg
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 8
(ng*hr/mL)/mg | 223 (105) | 103 (16.6) | 231 (110) | 204 (83.1) | 378 (110)
Statistical Analysis 1: Comparison: 1.0 mg/kg Antizol Followed by Ethanol vs Ethanol Followed by 1.0 mg/kg Antizol vs 3.0 mg/kg Antizol Followed by Ethanol vs Ethanol Followed by 3.0 mg/kg Antizol vs 5.0 mg/kg Antizol Followed by Ethanol; 1.0 mg/kg Cohort, 3.0 mg/kg cohort, 5.0 mg/kg cohort; Test type: Superiority; p = 0.0023, ANOVA — Overall p-value testing cohort difference from ANOVA
Statistical Analysis 2: Comparison: 1.0 mg/kg Antizol Followed by Ethanol vs Ethanol Followed by 1.0 mg/kg Antizol vs 3.0 mg/kg Antizol Followed by Ethanol vs Ethanol Followed by 3.0 mg/kg Antizol; 1.0 mg/kg Cohort, 3.0 mg/kg cohort; Test type: Superiority; p = 0.386, ANOVA — P-values for pairwise comparison between cohorts from ANOVA
Statistical Analysis 3: Comparison: 1.0 mg/kg Antizol Followed by Ethanol vs Ethanol Followed by 1.0 mg/kg Antizol vs 5.0 mg/kg Antizol Followed by Ethanol; 1.0 mg/kg, 5.0 mg/kg; Test type: Superiority; p = 0.0006, ANOVA — P-values for pairwise comparison between cohorts from ANOVA
Statistical Analysis 4: Comparison: 3.0 mg/kg Antizol Followed by Ethanol vs Ethanol Followed by 3.0 mg/kg Antizol vs 5.0 mg/kg Antizol Followed by Ethanol; 3.0 mg/kg, 5.0 mg/kg; Test type: Superiority; p = 0.0154, ANOVA — P-values for pairwise comparison between cohorts from ANOVA

7. Secondary Outcome: PK of 4-MP: AUC, From Time 0 Extrapolated to Infinite Time (AUC[0-∞])
Time Frame: as for outcome 2
Population: Modified Intent-to-Treat: participants who received any study medication or procedure, received study assessments through Study Day 2, and who had available data.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol
Number analyzed (Participants) | 1 | 2 | 1 | 1 | 6
ng*hr/mL | 11035 (NA) — 1 participant had an assessment | 7627 (948) | 55452 (NA) — 1 participant had an assessment | 57028 (NA) — 1 participant had an assessment | 136871 (43703)

8. Secondary Outcome: PK of 4-MP: DN AUC(0-∞)
Time Frame: as for outcome 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: (ng*hr/mL)/mg
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol
Number analyzed (Participants) | 1 | 2 | 1 | 1 | 6
(ng*hr/mL)/mg | 149 (NA) — 1 participant had an assessment | 122 (9.15) | 317 (NA) — 1 participant had an assessment | 334 (NA) — 1 participant had an assessment | 460 (129)

9. Secondary Outcome: PK of 4-MP: Percentage of AUC0-∞ Obtained by Extrapolation (AUC%Extrap)
Time Frame: as for outcome 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol
Number analyzed (Participants) | 1 | 2 | 1 | 1 | 6
percentage | 16.8 (NA) — 1 participant had an assessment | 13.0 (0.606) | 3.31 (NA) — 1 participant had an assessment | 4.37 (NA) — 1 participant had an assessment | 13.2 (12.6)

10. Secondary Outcome: PK of 4-MP: Half-Life (T1/2)
Time Frame: as for outcome 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol
Number analyzed (Participants) | 1 | 3 | 1 | 1 | 7
hours | 2.72 (NA) — 1 participant had an assessment | 3.11 (1.80) | 5.37 (NA) — 1 participant had an assessment | 5.76 (NA) — 1 participant had an assessment | 9.26 (4.93)

11. Secondary Outcome: PK of 4-MP: Apparent Clearance (CL/F)
Time Frame: as for outcome 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol
Number analyzed (Participants) | 1 | 2 | 1 | 1 | 6
L/hr | 6.70 (NA) — 1 participant had an assessment | 8.23 (0.618) | 3.15 (NA) — 1 participant had an assessment | 2.99 (NA) — 1 participant had an assessment | 2.35 (0.782)

12. Secondary Outcome: PK of 4-MP: Apparent Volume of Distribution During Terminal Phase (Vz/F)
Time Frame: as for outcome 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol
Number analyzed (Participants) | 1 | 2 | 1 | 1 | 6
Liters | 26.3 (NA) — 1 participant had an assessment | 24.7 (4.22) | 24.4 (NA) — 1 participant had an assessment | 24.9 (NA) — 1 participant had an assessment | 24.7 (9.91)

13. Secondary Outcome: PK of Ethanol: Cmax
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Placebo Followed by Ethanol: Placebo followed by ethanol 30 minutes later.
- Ethanol Followed by Placebo: Ethanol followed by placebo 30 minutes later.
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 8 | 24 | 8
mg/dL | 62.7 (10.1) | 70.3 (4.99) | 80.5 (5.20) | 43.3 (9.54) | 74.9 (21.9) | 59.3 (15.4) | 55.1 (14.5)
Statistical Analysis 1: Comparison: 1.0 mg/kg Antizol Followed by Ethanol; Test type: Superiority; ratio of parameter means = 115.57, 90% CI 2-sided [90.45 to 147.67] — Ratio of parameter means (Antizol/placebo, expressed as a percent), transformed back to the linear scale. 90% confidence interval for ratio of parameter means (expressed as a percent), transformed back to the linear scale
Statistical Analysis 2: Comparison: Ethanol Followed by 1.0 mg/kg Antizol; Test type: Superiority; ratio of parameter means = 126.05, 90% CI 2-sided [101.94 to 155.87] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: 3.0 mg/kg Antizol Followed by Ethanol; Test type: Superiority; ratio of parameter means = 137.58, 90% CI 2-sided [115.66 to 163.65] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: 3.0 mg/kg Antizol Followed by Ethanol; Test type: Superiority; ratio of parameter means = 82.4, 90% CI 2-sided [62.83 to 108.07] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: 5.0 mg/kg Antizol Followed by Ethanol; 3 participants in Cohort 3 had some residual 4-MP detected on Day 2 (Placebo treatment). As a result, the data for the participants on Day 2 were excluded from these statistical analyses, which could be compared with the analyses below where all available data were included; Test type: Superiority; ratio of parameter means = 115.25, 90% CI 2-sided [91.19 to 145.67] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: 5.0 mg/kg Antizol Followed by Ethanol; Analyses for Cohort 3 where all available data were included; Test type: Superiority; ratio of parameter means = 112.64, 90% CI 2-sided [96.14 to 131.98] — [estimate comment as in outcome 13, analysis 1]

14. Secondary Outcome: PK of Ethanol: DN Cmax
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: (mg/dL)/mg
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 8 | 24 | 8
(mg/dL)/mg | 0.00195 (0.000448) | 0.00198 (0.000420) | 0.00243 (0.000453) | 0.00155 (0.000359) | 0.00261 (0.000871) | 0.00193 (0.000667) | 0.00175 (0.000543)

15. Secondary Outcome: PK of Ethanol: Tmax
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 8 | 24 | 8
hours | 1.50 [0.500 to 2.50] | 0.833 [0.467 to 1.07] | 0.500 [0.500 to 0.500] | 1.42 [0.333 to 2.00] | 0.500 [0.333 to 1.50] | 0.500 [0.333 to 2.50] | 1.01 [0.833 to 2.00]

16. Secondary Outcome: PK of Ethanol: AUC(0-t)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 8 | 24 | 8
mg*hr/dL | 209 (46.1) | 209 (24.2) | 205 (13.1) | 135 (44.0) | 231 (67.1) | 157 (53.2) | 152 (42.6)
Statistical Analysis 1: Comparison: 1.0 mg/kg Antizol Followed by Ethanol; Test type: Superiority; ratio of parameter means = 139.63, 90% CI 2-sided [92.18 to 211.51] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Ethanol Followed by 1.0 mg/kg Antizol; Test type: Superiority; ratio of parameter means = 120.76, 90% CI 2-sided [108.80 to 134.03] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: 3.0 mg/kg Antizol Followed by Ethanol; Test type: Superiority; ratio of parameter means = 143.39, 90% CI 2-sided [107.72 to 190.87] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Ethanol Followed by 3.0 mg/kg Antizol; Test type: Superiority; ratio of parameter means = 103.13, 90% CI 2-sided [84.35 to 126.10] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: 5.0 mg/kg Antizol Followed by Ethanol; [analysis description as in outcome 13, analysis 5]; Test type: Superiority; ratio of parameter means = 123.17, 90% CI 2-sided [108.61 to 139.67] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: 5.0 mg/kg Antizol Followed by Ethanol; Analyses for Cohort 3 where all available data were included; Test type: Superiority; ratio of parameter means = 137.17, 90% CI 2-sided [123.30 to 152.59] — [estimate comment as in outcome 13, analysis 1]

17. Secondary Outcome: PK of Ethanol: DN AUC(0-t)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: (mg*hr/dL)/mg
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 8 | 24 | 8
(mg*hr/dL)/mg | 0.00648 (0.00171) | 0.00585 (0.00115) | 0.00613 (0.000641) | 0.00483 (0.00155) | 0.00791 (0.00163) | 0.00508 (0.00194) | 0.00476 (0.00124)

18. Secondary Outcome: PK of Ethanol: AUC(0-∞)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg*hr/mL
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 12 | 4 | 4 | 2 | 7 | 14 | 5
mg*hr/mL | 245 (55.7) | 263 (27.2) | 237 (27.0) | 215 (27.9) | 271 (75.0) | 214 (47.4) | 198 (47.3)
Statistical Analysis 1: Comparison: 1.0 mg/kg Antizol Followed by Ethanol; Test type: Superiority; ratio of parameter means = 121.81, 90% CI 2-sided [108.42 to 136.84] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Ethanol Followed by 1.0 mg/kg Antizol; Test type: Superiority; ratio of parameter means = 123.7, 90% CI 2-sided [93.55 to 163.56] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: 3.0 mg/kg Antizol Followed by Ethanol; Test type: Superiority; ratio of parameter means = 150.33, 90% CI 2-sided [93.14 to 242.63] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: 5.0 mg/kg Antizol Followed by Ethanol; Analysis for Cohort 3 where all available data were included; Test type: Superiority; ratio of parameter means = 122.83, 90% CI 2-sided [82.45 to 183.00] — [estimate comment as in outcome 13, analysis 1]

19. Secondary Outcome: PK of Ethanol: DN AUC(0-∞)
Time Frame: as for outcome 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: (mg*hr/dL)/mg
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 12 | 4 | 4 | 2 | 7 | 14 | 5
(mg*hr/dL)/mg | 0.00760 (0.00199) | 0.00731 (0.000843) | 0.00705 (0.000437) | 0.00768 (0.000707) | 0.00917 (0.00166) | 0.00681 (0.00182) | 0.00617 (0.00120)

20. Secondary Outcome: PK of Ethanol: AUC%Extrap
Time Frame: as for outcome 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 12 | 4 | 4 | 2 | 7 | 14 | 5
percentage | 14.7 (4.95) | 20.5 (6.90) | 13.2 (4.89) | 20.0 (4.68) | 12.1 (6.13) | 13.4 (5.62) | 13.9 (4.85)

21. Secondary Outcome: PK of Ethanol: T1/2
Time Frame: as for outcome 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 12 | 4 | 4 | 2 | 8 | 16 | 5
hours | 1.51 (0.391) | 1.95 (0.206) | 1.43 (0.219) | 1.78 (0.64) | 1.67 (0.608) | 1.45 (0.564) | 1.32 (0.193)

22. Secondary Outcome: PK of Ethanol: CL/F
Time Frame: as for outcome 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: dL/hr
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 12 | 4 | 4 | 2 | 7 | 14 | 5
dL/hr | 140 (36.8) | 138 (14.3) | 142 (8.81) | 131 (12.0) | 112 (19.6) | 159 (51.8) | 167 (32.7)

23. Secondary Outcome: PK of Ethanol: Vz/F
Time Frame: as for outcome 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: dL
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 12 | 4 | 4 | 2 | 7 | 14 | 5
dL | 297 (82.8) | 387 (57.0) | 295 (55.4) | 330 (89.5) | 242 (79.1) | 287 (86.3) | 321 (87.7)

24. Secondary Outcome: PK of Acetaldehyde: Cmax
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 8 | 24 | 8
µM | 59.6 (34.4) | 37.6 (26.9) | 50.9 (52.8) | 55.9 (52.2) | 40.0 (16.6) | 60.3 (34.8) | 42.7 (30.6)
Statistical Analysis 1: Comparison: 1.0 mg/kg Antizol Followed by Ethanol; Test type: Superiority; ratio of parameter means = 69.13, 90% CI 2-sided [48.88 to 97.78] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Ethanol Followed by 1.0 mg/kg Antizol; Test type: Superiority; ratio of parameter means = 124.46, 90% CI 2-sided [88.77 to 174.50] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: 3.0 mg/kg Antizol Followed by Ethanol; Test type: Superiority; ratio of parameter means = 105.31, 90% CI 2-sided [89.24 to 124.27] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Ethanol Followed by 3.0 mg/kg Antizol; Test type: Superiority; ratio of parameter means = 88.6, 90% CI 2-sided [56.66 to 138.54] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: 5.0 mg/kg Antizol Followed by Ethanol; [analysis description as in outcome 13, analysis 5]; Test type: Superiority; ratio of parameter means = 70.77, 90% CI 2-sided [34.16 to 146.59] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: 5.0 mg/kg Antizol Followed by Ethanol; Analyses for Cohort 3 where all available data were included; Test type: Superiority; ratio of parameter means = 86.04, 90% CI 2-sided [55.78 to 132.73] — [estimate comment as in outcome 13, analysis 1]

25. Secondary Outcome: PK of Acetaldehyde: DN Cmax
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µM/mg
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 8 | 24 | 8
µM/mg | 0.00181 (0.00101) | 0.00104 (0.000650) | 0.00157 (0.00167) | 0.00201 (0.00192) | 0.00138 (0.000542) | 0.00193 (0.00114) | 0.00141 (0.00112)

26. Secondary Outcome: PK of Acetaldehyde: Tmax
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 8 | 24 | 8
hours | 0.500 [0.167 to 5.50] | 0.650 [0.350 to 3.00] | 1.00 [0.333 to 3.50] | 1.33 [0.167 to 2.00] | 0.500 [0.333 to 2.50] | 0.500 [0.167 to 5.50] | 0.925 [0.167 to 4.00]

27. Secondary Outcome: PK of Acetaldehyde: AUC(0-t)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µM*hr
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 8 | 24 | 8
µM*hr | 178 (53.0) | 118 (56.4) | 155 (68.7) | 167 (84.4) | 128 (33.2) | 163 (61.3) | 139 (93.7)
Statistical Analysis 1: Comparison: 1.0 mg/kg Antizol Followed by Ethanol; Test type: Superiority; ratio of parameter means = 90.2, 90% CI 2-sided [69.54 to 117.00] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Ethanol Followed by 1.0 mg/kg Antizol; Test type: Superiority; ratio of parameter means = 112.28, 90% CI 2-sided [103.72 to 121.54] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: 3.0 mg/kg Antizol Followed by Ethanol; Test type: Superiority; ratio of parameter means = 106.08, 90% CI 2-sided [96.81 to 116.24] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Ethanol Followed by 3.0 mg/kg Antizol; Test type: Superiority; ratio of parameter means = 104.12, 90% CI 2-sided [83.50 to 129.84] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: 5.0 mg/kg Antizol Followed by Ethanol; [analysis description as in outcome 13, analysis 5]; Test type: Superiority; ratio of parameter means = 100.41, 90% CI 2-sided [77.86 to 129.49] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: 5.0 mg/kg Antizol Followed by Ethanol; Analyses for Cohort 3 where all available data were included; Test type: Superiority; ratio of parameter means = 94.7, 90% CI 2-sided [82.70 to 108.42] — [estimate comment as in outcome 13, analysis 1]

28. Secondary Outcome: PK of Acetaldehyde: DN AUC(0-t)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µM*hr/mg
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 8 | 24 | 8
µM*hr/mg | 0.00547 (0.00148) | 0.00329 (0.00144) | 0.00470 (0.00230) | 0.00597 (0.00293) | 0.00439 (0.00100) | 0.00521 (0.00204) | 0.00455 (0.00332)

29. Secondary Outcome: PK of Acetaldehyde: AUC(0-∞)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µM*hr
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 9 | 3 | 1 | 1 | 5 | 12 | 4
µM*hr | 234 (64.4) | 154 (63.3) | 297 (NA) — 1 participant had an assessment | 302 (NA) — 1 participant had an assessment | 188 (28.1) | 205 (71.1) | 227 (92.9)
Statistical Analysis 1: Comparison: 1.0 mg/kg Antizol Followed by Ethanol; Test type: Superiority; ratio of parameter means = 94.15, 90% CI 2-sided [78.01 to 1113.63] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: 5.0 mg/kg Antizol Followed by Ethanol; [analysis description as in outcome 13, analysis 5]; Test type: Superiority; ratio of parameter means = 107.05, 90% CI 2-sided [87.42 to 131.10] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: 5.0 mg/kg Antizol Followed by Ethanol; Analyses for Cohort 3 where all available data were included; Test type: Superiority; ratio of parameter means = 97.9, 90% CI 2-sided [84.84 to 112.97] — [estimate comment as in outcome 13, analysis 1]

30. Secondary Outcome: PK of Acetaldehyde: DN AUC(0-∞)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µM*hr/mg
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 9 | 3 | 1 | 1 | 5 | 12 | 4
µM*hr/mg | 0.00682 (0.00203) | 0.00432 (0.00176) | 0.00929 (NA) — 1 participant had an assessment | 0.0105 (NA) — 1 participant had an assessment | 0.00626 (0.00110) | 0.00616 (0.00171) | 0.00752 (0.00360)

31. Secondary Outcome: PK of Acetaldehyde: AUC%Extrap
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 9 | 3 | 1 | 1 | 5 | 12 | 4
percentage | 19.0 (6.07) | 18.8 (8.11) | 13.1 (NA) — 1 participant had an assessment | 9.78 (NA) — 1 participant had an assessment | 24.7 (5.26) | 13.7 (5.29) | 14.5 (11.4)

32. Secondary Outcome: PK of Acetaldehyde: T1/2
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 1.0 mg/kg Antizol | 3.0 mg/kg Antizol Followed by Ethanol | Ethanol Followed by 3.0 mg/kg Antizol | 5.0 mg/kg Antizol Followed by Ethanol | Placebo Followed by Ethanol | Ethanol Followed by Placebo
Number analyzed (Participants) | 10 | 3 | 1 | 1 | 6 | 12 | 4
hours | 3.14 (0.729) | 3.08 (0.640) | 2.48 (NA) — 1 participant had an assessment | 1.72 (NA) — 1 participant had an assessment | 3.45 (3.43) | 2.39 (0.521) | 2.09 (0.895)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from Check-In (Study Day 0) through Study Visit Day 7/Study End Visit
Groups:
- Pooled Placebo: Participants received placebo on either Study Day 1 or Study Day 2), administered 30 minutes prior to ethanol.
Arm/Group | Antizol 1.0 mg/kg | Antizol 3.0 mg/kg | Antizol 5.0 mg/kg | Pooled Placebo | Overall
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/8 | 0/8 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 13/16 | 6/8 | 8/8 | 21/32 | 28/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antizol 1.0 mg/kg (N=16) | Antizol 3.0 mg/kg (N=8) | Antizol 5.0 mg/kg (N=8) | Pooled Placebo (N=32) | Overall (N=32)
Headache (Nervous system disorders) | 5 | 1 | 3 | 7 | 15
Dysgeusia (Nervous system disorders) | 8 | 0 | 0 | 0 | 8
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 2 | 3
Blood pressure diastolic increased (Investigations) | 3 | 2 | 0 | 2 | 6
Blood pressure systolic decreased (Investigations) | 1 | 2 | 1 | 3 | 6
Respiratory rate increased (Investigations) | 6 | 0 | 5 | 5 | 15
Blood pressure systolic increased (Investigations) | 1 | 0 | 0 | 1 | 2
Tachycardia (Cardiac disorders) | 2 | 2 | 1 | 8 | 11
Bradycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 6 | 7
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 5 | 6
Blood LDH increased (Investigations) | 1 | 0 | 0 | 1 | 2 — lactic acid dehydrogenase (LDH)
Blood triglycerides increased (Investigations) | 0 | 1 | 0 | 1 | 2
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any Investigator/institution that plans on presenting or publishing results provide written notification of their request a minimum of 60 days prior to presentation or publication. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsors' Intellectual Property rights .